CLINICAL TRIAL: NCT03012243
Title: Randomized Controlled Trial of Bile Aspiration vs Drain in Acute Cholecystitis
Brief Title: Bile Aspiration vs Drain in Acute Cholecystitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bile aspiration vs drain trial
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cholecystitis, Acute
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Percutaneous Coronary Intervention; Cholecystostomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cholecystostomy (Active Comparator): Percutaneous cholecystostomy, leaving drain in situ
  Interventions: Procedure: Cholecystostomy
- Gallbladder aspiration (Experimental): Gallblader aspiration without drain
  Interventions: Procedure: Gallbladder aspiration

INTERVENTIONS:
Procedure: Gallbladder aspiration — Percutaneous ultrasound-guided aspiration of bile from the gallbladder. This is performed without leaving a drain in the gallbladder. The aspiration is performed with the intention to relief the pressure in the gallbladder, without drain.
  Other Names: Percutaneous intervention
  Arms: Gallbladder aspiration
Procedure: Cholecystostomy — Ultrasound-guided insertion of drain in the gallbladder. The drain is left in the gallbladder until clinical assessment and laboratory analyses show that the acute cholecystitis has been successfully treated.
  Other Names: Percutaneous intervention
  Arms: Cholecystostomy

SUMMARY:
In order to compare percutaneous cholecystostomy and leaving a drain in situ with percutaneous gallbladder aspiration we plan to undertake a double-blind randomized controlled trial.

DETAILED DESCRIPTION:
Percutaneous cholecystostomy is a minimally invasive technique for treatment of cholecystitis. The cholecystostomy can be inserted transhepatically or transabdominally. The transhepatic route is preferred due to lower risk for bile leakage. The drainage decompresses the gallbladder and drains the bile. This decompression reduces the inflammatory process in the gallbladder. Percutaneous cholecystostomy is often applied in patients not fit for emergency surgery who are in need of intervention due to deterioration of their clinical status. However, even though cholecystostomy is widely practised, it is not fully evaluated.

Percutaneous cholecystostomy has a high success rate, a low procedure-related mortality but a 30 day mortality of 15%. Furthermore, recurrence rates within one year after a cholecystostomy are reported to range between 4 to 22%.

The time duration of the drainage differ between different studies and range from three to six weeks. Optimal timing for drainage has not been studied. Two weeks seem to be sufficient for a maturation of the tract for the transhepatic route and 3 weeks for the transabdominal route. It has been suggested that a prolonged drainage duration is associated with increased risk for recurrence of inflammation due to local irritation of the gallbladder mucosa by the drain.

Percutaneous cholecystostomy is often considered as a bridge to surgery. However, less than half of patients treated with PC are treated with cholecystectomy. This suggests that this treatment is often chosen in a group not fit for surgery and often turns out to be a definitive treatment.

Percutaneous gallbladder aspiration is a technique used for purposes similar to percutaneous cholecystostomy. This technique is an alternative that may be more convenient than percutaneous cholecystostomy. The aspiration is performed with a small gauge needle under ultrasound guidance without leaving a drain. The aspiration leads to a decompression of the gallbladder, which facilitates recovery. However, it has only been described in a few studies and need more evaluation.

One single aspiration may be sufficient to relief symptoms for the majority of patients, but if two aspirations are performed the success rate increases substantially. One randomized controlled trial has been presented where PC is compared to gallbladder aspiration. In this trial PC was superior to gallbladder aspiration in terms of effectiveness. In this trail, however, only one aspiration was performed. No major complications occurred in either group and minor complications were equal between the groups. In a retrospective study comparing aspiration with PC it was found that gallbladder aspiration is safer than PC and has a comparable clinical outcome.

It is believed that single decompressions are sufficient for reduction of the intraluminal pressure. Only a minority of patients have positive bile cultures which, indicates that infection is not a key mechanism in development of cholecystitis, which indicates that a continuous drainage may not be necessary. As lower rates of complications are reported for aspiration due to usage of smaller needle and no drain left that can dislocate and cause bile leakage which is feared complication of PC. It is suggested that PC can have a role as a salvage method when aspiration is not successful.

In order to compare percutaneous cholecystostomy and leaving a drain in situ with percutaneous gallbladder aspiration we plan to undertake a double-blind randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Acute cholecystitis, not warranting acute cholecystectomy

Exclusion Criteria:

* Indication for acute cholecystectomy, i.e. history < 5 days and no contraindication to surgery
* Liver cirrhosis
* Ascites
* Emphysematous cholecystitis
* Gallbladder perforation
* Suspected malignant condition
* Portal Hypertension
* Biliary pancreatitis
* Common bile duct stones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Amount of morphine administrated | 24 hours
  The total amount of morphine required to relieve the pain the first 24 hours

SECONDARY OUTCOMES:
Pain | 5 days
  Pain intensity rated on a Visual Analogue Scale
Nausea | 5 days
  Nausea estimated with a Likert scale
Re-intervention | 5 days
  Repeated percutaneous aspiration of adjustment of drain
Body temperature | 5 days
  Temperature measured daily
CRP | 5 days
  Daily measures of C-reactive protein
LPK | 5 days
  Daily measures of Leukocyte particle Concentration
Time to discharge | 30 days
  Time from intervention to discharge from the hospital
Complications | 30 days
  Procedure-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Sandblom, Assoc Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Center for Digestive Diseases, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No